CLINICAL TRIAL: NCT07055152
Title: Retinal OCTA for Microvascular Dysfunction Evaluation and Outcome Prediction in MINOCA Patients
Acronym: REVEAL
Status: Recruiting | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Mattia Alberti, Principal Investigator, University of Pisa
Other Study IDs: REVEAL
Record Dates: First submitted 2025-06-19; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: MINOCA; STEMI; Normal
MeSH Terms: conditions — MINOCA; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MINOCA: MINOCA
- STEMI: STEMI
- NORMAL: NORMAL

SUMMARY:
The aim of this study is to evaluate microvascular dysfunction through OCTA in MINOCA patients. In order to better understand the condition, OCTA will also be performed in two matched patient groups: healthy controls and ACS patients. The study will compare the retinal microvascular parameters across these groups to determine differences in microvascular function in MINOCA patients. Additionally, in the MINOCA subgroup, the study will further evaluate the differences in microvascular dysfunction within specific subsets of patients (e.g., Takotsubo, vasospastic angina, microvascular angina, patients with evidence of plaque erosion) to understand the variability and potential mechanisms underlying each subgroup of MINOCA.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients aged > 18.

Diagnosis:

MINOCA Group: Patients diagnosed with Myocardial Infarction with Non-Obstructive Coronary Arteries (MINOCA) confirmed by coronary angiography.

ACS Group: Patients with Acute Coronary Syndrome (ACS) with significant coronary artery stenosis which are matched with MINOCA patients for gender, age, LVEF at admission and chronic kidney disease stage.

Healthy Controls: Age and gender-matched healthy individuals with no history of cardiovascular disease.

Consent: Written informed consent obtained from all participants. Feasibility: Ability to undergo OCTA and other required imaging procedures.

Exclusion Criteria:

* Ocular Conditions: Any significant ocular disease (e.g., glaucoma, diabetic retinopathy, macular degeneration) that could interfere with OCTA imaging quality.

Severe Comorbidities: Presence of severe systemic diseases, such as advanced renal failure, active cancer, or severe liver disease, which might impact study participation.

Coronary Artery Disease or Myocarditis: For the MINOCA group, patients with coronary artery stenosis > 50% or functionally significant (FFR <0.8) or patients with Myocarditis detected through CMR will be excluded Pregnancy: Pregnant or breastfeeding women. Inability to Comply: Patients unable or unwilling to comply with study procedures, including follow-up visits.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: MINOCA Group: Patients diagnosed with Myocardial Infarction with Non-Obstructive Coronary Arteries (MINOCA) confirmed by coronary angiography.
  ACS Group: Patients with Acute Coronary Syndrome (ACS) with significant coronary artery stenosis which are matched with MINOCA patients for gender, age, LVEF at admission and chronic kidney disease stage.
  Healthy Controls: Age and gender-matched healthy individuals with no history of cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
OCTA changes in three different courts and their correlation with clinical and imaging biomarkers | 24 months
  ETDRS Grid Parameters: The macular area will be divided into the following regions for detailed analysis:
  Central (Foveal) Zone Inner Ring (split into quadrants: superior, inferior, nasal, temporal) Outer Ring (split into quadrants: superior, inferior, nasal, temporal)
  Foveal Avascular Zone (FAZ): The following characteristics will be recorded:
  FAZ Area (mm^2) FAZ Perimeter (mm) FAZ Circularity Index

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pisa, Cisanello Hospital, Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Shared upon reasonable requests